CLINICAL TRIAL: NCT01126944
Title: Study of Congestive Heart Failure Through the Evaluation of Cardiac Resynchronization Non-responders and Mechanical Assistance Therapy
Brief Title: LVAD in Non Cardiac Transplant Candidates and Non Responders to Resynchronization
Acronym: CHECKMATE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients recruted since recruiting is open
Sponsor: Rennes University Hospital (Other)
Collaborators: Thoratec Europe Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOC/09-03
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2010-09

CONDITIONS: Heart Failure at NYHA Stage III or IV; Non Responders to Resynchronization; Non Candidates for Transplantation
Keywords: heart failure; resynchronization; left ventricular assist device
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- system heart mate II (Experimental): left ventricular assist device
  Interventions: Device: heart mate II
- normal medical care (No Intervention): Optimal medical treatment for heart failure according to international guidelines

INTERVENTIONS:
Device: heart mate II — left ventricular assist device
  Arms: system heart mate II

SUMMARY:
The prognosis for heart failure patients is bleak for the advanced stages of the disease, with a reported 6-month mortality rate of almost 50% in patients treated with chronic inotropic therapy. As well as its very severe prognosis, heart failure is a costly disease. Heart transplantation remains the reference treatment for the terminal stage of the disease but although this is an effective therapy, it does engender ethical, social, economic and legal problems. It also requires irreproachable and costly logistics, immuno-suppressor treatment and a lifetime of follow-ups. In particular, the number of donors has been going down steadily for several years in most countries which offer a heart transplant programme and some patients cannot take advantage of being added to a waiting list for a graft (age, co-morbidities…).

It is in this context that, alongside the medical treatments for cardiac insufficiency, other therapeutic strategies were developed, including resynchronization and long-term mechanical circulatory support. The progress made in resynchronization is at several levels: better understanding of the action mechanisms, the development and improvement of equipment specifically dedicated to resynchronization and prospective and randomized clinical trials which have scientifically validated this technique.

Simultaneously, many studies were published evaluating long term support with mechanical circulatory support (MCS), excluding light devices, as a bridge to transplant or an alternative to a transplant. It is also recognized that mechanical circulatory support with a new generation of continuous flow assist device improved the quality of life and functional capacity, with a reduced risk of device failure and infrequent need for replacement.

The "Achilles heel" of cardiac resynchronization remains the 20 to 40% of patients who respond barely or not at all. Among this population of patients, some are not candidates for a transplantation and long-term mechanical circulatory support by axial pump is an alternative to be considered. We elaborated an original randomized pilot study for these patients in order to evaluate their survival and their quality of life, to define if they should be proposed a left ventricular assist device (LVAD)or not.

ELIGIBILITY:
Inclusion Criteria:

* patients with heart failure class III or IV NYHA
* LVEF < 35%
* resynchronization for at least 6 months
* non eligibility for cardiac transplant
* operability and psychological criteria assessed

Exclusion Criteria:

* Patients incapable of understanding the proposed procedure, its risks and potential benefits or the consequences engendered by the permanent implanting of a left ventricular assist device
* Patients on mechanical circulatory support, including an intra-aortic counter-pulsion balloon, at the time of randomisation
* Patients with acute decompensated cardiac insufficiency at the time of randomisation
* Patients whose body surface area is below 1.2m²
* Patients with a mechanical cardiac valve
* Patients requiring associated aortic or mitral surgery
* Patients with an active uncontrolled infection
* Patients with a severe pulmonary respiratory pathology
* Patients with contra-indications for or an intolerance to anti-coagulants or platelet anti-aggregants
* Presence of risk factors or indicators of visceral failure (severe COPD, renal insufficiency with dialysis, hepatic insufficiency with cholestasis…)
* Patients with a Lietz/Miller operating mortality score ≥ "high risk"
* Patients with an elevated risk of an embolism and atrial intra-cardiac thrombus
* Severe right ventricular failure (echography and right cardiac catheter examination) with the probable need for right ventricular mechanical assistance
* Patients who are candidates for coronary revascularisation
* Participation in another study which may interact with the proposed clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
quality of life : minnesota living with heart failure | one year

SECONDARY OUTCOMES:
6 mn walk test | one year

CONTACTS AND LOCATIONS:
Locations (4):
- France (3):
  - La Timone Hospital, Marseille
  - La Pitié Salpétrière Hospital, Paris
  - University Hospital, Rennes
- Klinik für Herz- und Thoraxchirurgie Martin-Luther-Universität, Halle, Germany